CLINICAL TRIAL: NCT00474695
Title: VEGF and HTRA1 DNA Polymorphisms in Neovascular AMD Pathogenesis and Response to Lucentis
Brief Title: Study Evaluating Genotypes Using Lucentis
Acronym: SEAGUL
Status: Terminated | Type: Observational
Why Stopped: IND holder relocated from the University of Utah
Sponsor: University of Utah (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Paul S. Bernstein, Professor, Ophthalmology, University of Utah
Other Study IDs: 21441; SEAGUL
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Age-Related Maculopathy
Keywords: Exudative age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Active approved treatment
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Lucentis — 0.05 mg intravitreal injection
  Other Names: ranibizumab

SUMMARY:
The purpose of the study is to investigate whether the efficacy of Lucentis treatment for exudative age-related macular degeneration is associated with VEGF and HTRA1 DNA polymorphisms

DETAILED DESCRIPTION:
Treatment naive exudative AMD patients will receive Lucentis treatment as standard of care, and followed monthly for 12 months. Standard ophthalmologic exams will be performed, along with ETDRS visual acuity and optical coherence tomography (OCT). A blood sample will be obtained for DNA analysis. The primary outcome measure is change in visual acuity at 4 months after initial Lucentis treatment. Secondary outcomes are change in visual acuity and retinal thickness at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive AMD patients;
* At least 50 years of age;
* Visual acuity between 20/40 and 20/320

Exclusion Criteria:

* Pregnancy;
* Prior enrollment in a ranibizumab clinical trial;
* Previous therapy in either eye for AMD;
* Concurrent eye disease that could compromise visual acuity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moran Eye Center Clinic
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the VEGF and HTRA1 genotypes associated with improvement in visual acuity | 4 months

SECONDARY OUTCOMES:
Determine VEGF and HTRA1 genotypes associated with change or no change in visual acuity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bernstein, MD, PhD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - California Retina Consultants, Santa Barbara, California
  - Porter Adventist Hospital, Denver, Colorado
  - University of Utah, Moran Eye Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Zhao L, Grob S, Avery R, Kimura A, Pieramici D, Lee J, Rabena M, Ortiz S, Quach J, Cao G, Luo H, Zhang M, Pei M, Song Y, Tornambe P, Goldbaum M, Ferreyra H, Kozak I, Zhang K. Common variant in VEGFA and response to anti-VEGF therapy for neovascular age-related macular degeneration. Curr Mol Med. 2013 Jul;13(6):929-34. doi: 10.2174/15665240113139990048. PMID 23745581